CLINICAL TRIAL: NCT03555799
Title: Evaluation of Changes of Venous Return After Spinal and Epidural Analgesia and Anesthesia by Ultrasound Guided Vena Cava Diameter Measurement
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Other Study IDs: 1194575
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy Related; Hypotension, Orthostatic
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Labor analgesia patients: Patients with clinical indication of labor epidural will have IVC diameter measurement with ultrasound before and after the epidural placement
  Interventions: Diagnostic Test: Inferior vena cava ultrasound

INTERVENTIONS:
Diagnostic Test: Inferior vena cava ultrasound — Abdominal ultrasound to identify IVC between hepatic veins and right atrium. Measurement of dimensions throughout respiratory cycle (before and after labor epidural)

SUMMARY:
The investigators propose this study to test the hypotheses that inferior vena cava (IVC) diameter can predict hypotension after labor analgesia (epidural, combined spinal-epidural) and neuraxial anesthesia for cesarean section (epidural, combined spinal-epidural and spinal block) in full-term pregnant patients.

DETAILED DESCRIPTION:
After approval by the Institutional Review Board and patient consent, term pregnant patients (>37 week gestation) admitted to the obstetric service of Augusta University Medical Center, who require administration of neuraxial analgesia for labor or regional anesthesia for cesarean section, will be included in the study. The consent will be obtained by the attending, resident or medical student in which the investigators will explain to the patient the procedure, benefit, risk, cost and, confidentiality. The investigators plan to get the consent immediately after the patient arrived at the unit to avoid any interference with the delivery process. If the patient needs to go to an emergency cesarean section. This patient is not going to be included in the study. Demographic variables (age, BMI, Gravity, parity and gestation weeks) and hemodynamic variables (MAP and HR) will be recorded. All patients will be lying in supine position, breathing spontaneously. The ultrasound examination will be performed before commencement of the neuraxial procedure and will be repeated two minutes after administration of the neuraxial anesthetic. Ultrasound measurements will be made with a Sonosite Edge (Sonosite Inc. USA) machine and a C60X curved linear phased array transducer (Sonosite Inc.) set to abdominal mode. All measurements will be made by two attending anesthesiologists (ERP and AR) who have experience in transthoracic echocardiography, and a resident who receives the basic instruction to measure IVC diameter. The medical student will be present during the procedure and will ensure that the study echocardiographic views are taken.

The IVC will be visualized using a paramedian long-axis view via a subcostal approach according to guidelines of the American Society of Echocardiography. A two-dimensional image of the IVC will be obtained and pulsed wave Doppler will be used to differentiate from the aorta. Variations in IVC diameters will be assessed with M-mode applied 2 cm. distal to the right atrium. To ensure consistent measurements, each operator will take three images. The best quality images are chosen. Maximum and minimum IVC diameters during a single respiratory cycle will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients >37 weeks of gestation
2. Indication for neuraxial labor analgesia or regional anesthesia for cesarean section
3. Age older than 18 years
4. Pregnancy without diagnosed comorbidities

Exclusion criteria:

1. Unwillingness to participate in the study
2. Diagnosis of Hypertensive disorders of pregnancy
3. Diagnosis of cardiopulmonary disease
4. Allergy to US gel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Parturients in labor
Study Population: Term pregnant patients in labor who have labor epidural placement.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
IVC diameter | 10 minutes
  IVC diameter in centimeters during respiratory cycle

SECONDARY OUTCOMES:
Mean arterial pressure | 30 minutes
  Mean arterial pressure
Nausea | 30 minutes
  Nausea

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No